CLINICAL TRIAL: NCT07176338
Title: Lens Epithelial Cell Proliferation in Patients Suffering From Diabetes and Treated With Metformin in Vitro: a Pilot Study
Brief Title: Role of Metformin in Posterior Capsule Opacification
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PCO Metformin
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cataract; Diabetes Mellitus Type 2
MeSH Terms: conditions — Cataract; Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin Concentration in Blood Serum and Lens capsule (Experimental)
  Interventions: Diagnostic Test: Blood and lens capsule samples for PK testing

INTERVENTIONS:
Diagnostic Test: Blood and lens capsule samples for PK testing — Blood samples and lens capsule tissue will be collected from patients for PK testing

SUMMARY:
Determination of concentrations of systemically applied metformin in human lens capsule and its ability to lower the proliferation rate of human lens epithelial cells in vitro.

DETAILED DESCRIPTION:
Cataract remains a leading cause of visual impairment and blindness worldwide, particularly in aging populations. Although several pharmacological approaches have been explored, removal of the lens with phacoemulsification remains the gold standard of treatment. This surgical technique removes the opacified lens while preserving the capsular bag to hold an intraocular lens (IOL).

Despite its overall safety and efficacy, cataract surgery is frequently complicated by posterior capsule opacification (PCO), the most common long-term postoperative issue. PCO leads to secondary visual deterioration and is observed in approximately 20-30% of patients within five years of surgery. The standard treatment for visually significant PCO is neodymium-doped yttrium-aluminium-garnet (Nd:YAG) laser capsulotomy, a rapid and effective outpatient procedure, though not without risks such as increased intraocular pressure, cystoid macular edema, or retinal detachment.

The pathophysiology of PCO involves residual lens epithelial cells (LECs) proliferating, migrating, and undergoing epithelial-mesenchymal transition (EMT), ultimately leading to fibrotic or regenerative capsular changes. Fibrotic variants are characterized by matrix contraction and EMT, while regenerative types manifest as Elschnig pearls.

Multiple risk factors have been associated with PCO, including age, ocular inflammation, and systemic diseases. However, the current evidence remains inconsistent: some studies suggest diabetes may exert a protective effect against PCO, whereas others report an increased risk with longer disease duration. These discrepancies may be due to the lack of subgroup analyses with respect to antidiabetic therapy. In particular, metformin use might act as a protective factor, whereas diabetes without metformin treatment could increase PCO risk. The absence of stratification by medication may thus explain the heterogeneous findings. Beyond PCO, diabetes is linked to multiple ocular comorbidities including retinopathy, ocular surface disease, and a higher overall risk for cataract formation.

Metformin is the most widely prescribed oral antidiabetic drug and exerts pleiotropic effects beyond glucose control. It has demonstrated antifibrotic, antiproliferative, and anti-senescent properties in various tissues. Preclinical studies indicate that metformin suppresses LEC senescence and proliferation, and recent clinical data link metformin use to reduced rates of Nd:YAG laser capsulotomy. In systemic contexts, metformin modulates fibrotic and proliferative responses in hepatic, renal, cardiovascular, and neoplastic tissues primarily via activation of AMP-activated protein kinase (AMPK), inhibition of mTOR signaling, and reduction of oxidative stress and inflammatory pathways.

While metformin has been detected in aqueous humour, its presence and concentration in the human lens capsule remain unknown. Moreover, it is unclear whether intraocular metformin levels are sufficient to affect LEC proliferation-an essential driver of PCO pathogenesis. Previous studies have not established a link between systemic metformin exposure and functional intraocular bioactivity, nor have they used live-cell tracking to directly assess it's effect on LEC behaviour.

In addition to systemic and pharmacological factors, IOL design also influences PCO development. A sharp square-edge design acts as a mechanical barrier to LEC migration and remains the current standard in PCO prevention. Hydrophobic acrylic materials are associated with lower PCO rates compared to hydrophilic or polymethylmethacrylate (PMMA) optics, although none completely prevent it.

Therefore, the aim of the study is to quantify metformin concentrations in serum and lens capsule tissue of type 2 diabetes mellitus patients and to assess the effect of metformin on human LEC proliferation in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Diabetes mellitus type II
* Metformin treatment
* Age 21 or older
* Written informed consent prior to surgery

Exclusion Criteria:

* Diabetes mellitus type I
* Previous ocular surgery or trauma regarding cataract surgery
* Previous vitrectomy
* Pregnancy (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Metformin concentration in the human lens capsule | 12 months

SECONDARY OUTCOMES:
Metformin concentration in human blood | 12 months
Influence of Metformin on in vitro proliferation of LECs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS)
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided